CLINICAL TRIAL: NCT02998957
Title: Efficacy of Transcutaneous Electrical Stimulation at Dingchuan (EX-B1) in Hospitalized COPD Patients With Severe Dyspnoea: Patient and Assessor Blinded Randomized Placebo Control Trial
Brief Title: Acupoint Transcutaneous Electrical Nerve Stimulation in Hospitalized COPD Patients With Severe Dyspnoea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIC-195-15
Record Dates: First submitted 2016-11-30; First posted 2016-12-21 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Acupuncture; TENS; Physiotherapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AcuTENS (Experimental): Stimulation using a portable TENS electrostimulation device at Dingchuan point using a biphasic rectangular wave with a frequency of 2Hz and a pulse width of 200 ms. The stimulation will be achieved using the highest intensity tolerated by the patient without pain during 40 minuts.
  Once a day during 5 consecutive days.
  Interventions: Device: AcuTENS
- Sham AcuTENS (Sham Comparator): Stimulation using a modified portable TENS electrostimulation device at Dingchuan point with no electrical output, even though the screen will light up and display the same data as in the unmodified device during 40 minuts. Patients in this group will be informed that, due to the frequency of stimulation, it is unlikely that they will feel the electric stimulation.
  Once a day during 5 consecutive days.
  Interventions: Device: Sham AcuTENS

INTERVENTIONS:
Device: AcuTENS — Stimulation of acupuncture point Dingchuan using transcutaneous electrical nerve stimulation (TENS) instead of needles
  Other Names: TENS; Acupoint transcutaneous electrical nerve stimulation
  Arms: AcuTENS
Device: Sham AcuTENS — Portable TENS electrostimulation device with no electrical output
  Arms: Sham AcuTENS

SUMMARY:
Introduction:

Chronic obstructive pulmonary disease (COPD) presents with a gradual reduction and little bitterness reversible airflow causing shortness of breath, chronic cough and sputum abnormal. Patients with COPD often suffer exacerbations of their symptoms, particularly dyspnea, causing hospital admissions. Recent studies have shown that acupuncture stimulation transcutánea (AcuTENS) Dingchuan point (EX-B1) could help reduce dyspnea in patients with COPD.

Objective:

The aim of this study was to evaluate the possible utility of adding to the usual treatment stimulation AcuTENS in COPD patients admitted with severe dyspnea.

Methodology:

Patients who agree to participate will be randomly divided into two groups. The intervention group will receive a daily treatment, during the period of hospitalization, 45 minutes stimulation at acupuncture point AcuTENS Dingchuan (EX-B1), while the control group performed the same procedure with a device TENS simulated. The extent of dyspnea in both groups as well as the number of days of hospitalization and the number of drugs consumed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 45 and 70 years, with a diagnose of COPD according to the GOLD guidelines.
2. Patients with one episode of hospitalization for COPD exacerbation in the past year, but not more than three episodes.
3. Smoking habit history of more than 10 packages-year.
4. Patients able to correctly understand and answer the modified Borg scale.
5. Patiens with an initial degree of dyspnoea with a score of at least 5 in the modified Borg scale.
6. Patients recruited for the study during the first 48 hours of their hospitalization.
7. Patients who accept to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Patients with any contraindication for transcutaneous electrical stimulation (patiens with pacemakers, skin injury in the application area ...).
2. Patiens with any cardiovascular, neurological or psychiatric disease that may affect the perception of dyspnea.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Dyspnoea | At baseline, day 1, day 2, day 3 day 4 and day 5 of the study.
  Change from baseline using the modified Borg scale

SECONDARY OUTCOMES:
Hospitalization days | Up to 1 months after discharge
  Number of days from the time of admission until discharge will be collected from the patient's clinical history
Quantity of drug administered | Up to 1 months after discharge
  Amount of drugs administered during the hospitalization will be determined by data collected from the patient's clinical history
Peak expiratory flow | At baseline, day 1, day 2, day 3 day 4 and day 5 of the study.
  Change from baseline using a peak flow meter
PaO2 | At baseline, day 1, day 2, day 3 day 4 and day 5 of the study. (only if there is a medical indication for it)
Mortality | Up to 3 months after discharge
  Percentage of deaths 3 months after discharge
PaCO2 | At baseline, day 1, day 2, day 3 day 4 and day 5 of the study. (only if there is a medical indication for it)
Arterial blood pH | At baseline, day 1, day 2, day 3 day 4 and day 5 of the study. (only if there is a medical indication for it)
SaO2 | At baseline, day 1, day 2, day 3 day 4 and day 5 of the study. (only if there is a medical indication for it)
Relapses | Up to 3 months after discharge
  Percentage of relapses 3 months after discharge
Readmissions | Up to 3 months after discharge
  Percentage of readmissions 3 months after discharge

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Sant Joan de Déu de Manresa, Manresa, Barcelona
  - Parc Sanitari de Sant Joan de Déu, Sant Boi de Llobregat, Barcelona
  - Hospital del Mar, Barcelona